CLINICAL TRIAL: NCT00900276
Title: BARC: A Secreted Marker of Kidney Cancer
Brief Title: Biomarkers in Patients With Kidney Cancer or Cancer of the Urothelium and in Healthy Participants
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00000577; P30CA012197 (NIH); CCCWFU-89A06; CCCWFU-IRB00000577
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Bladder Cancer; Kidney Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: localized transitional cell cancer of the renal pelvis and ureter; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder; stage I renal cell cancer; stage II renal cell cancer; recurrent renal cell cancer; recurrent bladder cancer; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; anterior urethral cancer; posterior urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Kidney Neoplasms; Urethral Neoplasms; Carcinoma, Renal Cell | interventions — Immunologic Techniques; Mass Spectrometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: immunologic technique
Other: laboratory biomarker analysis
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood and urine from patients with cancer and from healthy participants in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This laboratory study is looking at biomarkers in patients with kidney cancer or cancer of the urothelium and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether bone morphogenetic protein antagonist regulated in cancer (BARC) is present in urine and serum samples from patients with renal cell carcinoma or transitional cell carcinoma of the urothelium and from healthy participants and whether changes in BARC expression levels in these fluids correlate with various disease states.
* Evaluate BARC's utility as a biomarker of kidney cancer.
* Determine whether differences in BARC levels exist between patients with cancer vs non-cancer patients visiting the urology clinic.
* Determine whether differences in BARC levels exist among the different types of kidney cancers.
* Evaluate serum markers of iron metabolism and determine whether changes in BARC expression correlates with changes in these systemic iron markers.
* Determine whether the development of an enzyme-linked immunosorbent assay to detect BARC levels as a diagnostic procedure is feasible and desirable.

OUTLINE: This is a pilot study.

Blood and urine samples are collected. Samples are evaluated by immunoblotting to detect bone morphogenetic protein antagonist regulated in cancer (BARC) and by mass spectrometry analysis to detect hepcidin levels. Serum samples are further analyzed for serum iron, ferritin, and total-iron body capacity. Histology of biopsy samples will be recorded for patients undergoing nephrectomy for renal cell carcinoma. These patients will undergo a second collection of blood and urine samples 3 months post-nephrectomy.

ELIGIBILITY:
Inclusion:

* Age > 18 years
* Meets 1 of the following criteria:

  * Diagnosis of renal cell carcinoma, meeting all of the following criteria:

    * Suitable surgical candidate
    * No clinical or pathologic T stage > T2
    * No clinical or pathologic evidence of vein and/or lymph node involvement
    * No evidence of metastatic disease as evaluated by abdominal/pelvic CT scan or MRI, chest x-ray or chest CT scan, and bone scan (if alkaline phosphatase abnormal)
  * Diagnosis of transitional cell carcinoma of the urothelium

    * Currently undergoing Bacille calmette-guérin (BCG) therapy OR has not received prior BCG therapy
  * Healthy participant (control)

    * No history of carcinoma

Exclusion:

* Previous or concurrent malignancy except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* Serious medical or psychiatric illness that would preclude study compliance
* Current participation in a treatment related research study within the last 30 days
* Acute illness
* Bleeding disorder or dyscrasia

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those with a diagnosis of renal cell carcinoma or a diagnosis of transitional cell carcinoma of the urothelium.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Presence of bone morphogenetic protein antagonist regulated in cancer (BARC) in urine and serum samples
BARC expression levels
Correlation of changes in serum markers of iron metabolism with changes in BARC expression
Feasibility of an enzyme-linked immunosorbent assay to detect BARC levels as a diagnostic procedure

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Torti, MD, MPH, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States